CLINICAL TRIAL: NCT00092742
Title: A Randomized, Double-Blind, Multicenter Study to Evaluate the Tolerability and Effectiveness of Etoricoxib 90 mg q.d. vs. Diclofenac Sodium 75 mg b.i.d. in Patients With Rheumatoid Arthritis
Brief Title: Investigational Drug Versus an Approved Drug in Patients With Rheumatoid Arthritis (0663-072)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-072; 2004_055
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Arcoxia
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663, etoricoxib
Drug: Comparator: Diclofenac sodium

SUMMARY:
The purpose of this study is to evaluate the long-term safety of an investigational drug versus an approved drug for the relief of pain in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
The duration of treatment is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 50 years or older with rheumatoid arthritis.

Exclusion Criteria:

* History of gastrointestinal malabsorption or inflammatory bowel disease
* History of heart problems such as: congestive heart failure (CHF), heart attack or high blood pressure.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4086 (Actual)
Dates: Start 2003-02; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Discontinuations due to clinical and laboratory gastrointestinal adverse experiences

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Cannon CP, Curtis SP, FitzGerald GA, Krum H, Kaur A, Bolognese JA, Reicin AS, Bombardier C, Weinblatt ME, van der Heijde D, Erdmann E, Laine L; MEDAL Steering Committee. Cardiovascular outcomes with etoricoxib and diclofenac in patients with osteoarthritis and rheumatoid arthritis in the Multinational Etoricoxib and Diclofenac Arthritis Long-term (MEDAL) programme: a randomised comparison. Lancet. 2006 Nov 18;368(9549):1771-81. doi: 10.1016/S0140-6736(06)69666-9. PMID 17113426
- [Background] Krueger K, Lino L, Dore R, Radominski S, Zhang Y, Kaur A, Simpson R, Curtis S. Gastrointestinal tolerability of etoricoxib in rheumatoid arthritis patients: results of the etoricoxib vs diclofenac sodium gastrointestinal tolerability and effectiveness trial (EDGE-II). Ann Rheum Dis. 2008 Mar;67(3):315-22. doi: 10.1136/ard.2007.082388. Epub 2007 Oct 27. PMID 17965424
- [Background] Krum H, Curtis SP, Kaur A, Wang H, Smugar SS, Weir MR, Laine L, Brater DC, Cannon CP. Baseline factors associated with congestive heart failure in patients receiving etoricoxib or diclofenac: multivariate analysis of the MEDAL program. Eur J Heart Fail. 2009 Jun;11(6):542-50. doi: 10.1093/eurjhf/hfp054. Epub 2009 Apr 19. PMID 19380329
- [Background] Laine L, Curtis SP, Langman M, Jensen DM, Cryer B, Kaur A, Cannon CP. Lower gastrointestinal events in a double-blind trial of the cyclo-oxygenase-2 selective inhibitor etoricoxib and the traditional nonsteroidal anti-inflammatory drug diclofenac. Gastroenterology. 2008 Nov;135(5):1517-25. doi: 10.1053/j.gastro.2008.07.067. Epub 2008 Aug 3. PMID 18823986
- [Background] Laine L, Goldkind L, Curtis SP, Connors LG, Yanqiong Z, Cannon CP. How common is diclofenac-associated liver injury? Analysis of 17,289 arthritis patients in a long-term prospective clinical trial. Am J Gastroenterol. 2009 Feb;104(2):356-62. doi: 10.1038/ajg.2008.149. Epub 2009 Jan 27. PMID 19174782